CLINICAL TRIAL: NCT06909994
Title: Sensory Function and Its Relationship With Motor Performance and Daily Living Activities in Young Adults With Cerebral Palsy
Brief Title: Daily Living Activities in Young Adults With Cerebral Palsy
Acronym: Palsy202503
Status: Completed | Type: Observational
Sponsor: Universidad de Burgos (Other)
Responsible Party: Sponsor
Other Study IDs: Palsy202503; UBurgos (Other: Universidad de Burgos)
Record Dates: First submitted 2025-03-26; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy; Sensitivity; Motor Skills Disorders; Activity, Motor
MeSH Terms: conditions — Cerebral Palsy; Hypersensitivity; Motor Skills Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Young Adults: A multicenter cross-sectional study was conducted involving two groups of 36 participants aged 16-45 years. Sensory and motor variables were assessed using the Semmes-Weinstein Monofilaments, Two-Point Discrimination Test, Modified Ashworth Scale, Digital Dynamometer, Box and Block Test, Functional Independence Measure, and the Lawton and Brody Scale.
- Cerebral Palsy: A multicenter cross-sectional study was conducted involving two groups of 36 participants aged 16-45 years. Sensory and motor variables were assessed using the Semmes-Weinstein Monofilaments, Two-Point Discrimination Test, Modified Ashworth Scale, Digital Dynamometer, Box and Block Test, Functional Independence Measure, and the Lawton and Brody Scale.
  Interventions: Other: individual assessments

INTERVENTIONS:
Other: individual assessments — Participants in the CP group underwent individual assessments using seven standardized instruments to evaluate sensory and motor function, as well as independence in daily activities. Data collection was conducted in person at the participating institutions by trained professionals following a structured protocol. All procedures were performed after verifying cognitive eligibility (score ≥ 19) and obtaining informed consent. The same protocol was applied across both centers to ensure consistency. The control group followed the same assessment process. Each evaluation session lasted approximately two hours per participant.
  Groups: Cerebral Palsy

SUMMARY:
This study explored the relationship between sensory function and occupational performance in young adults with Cerebral Palsy. Using standardized assessments, researchers compared tactile sensitivity and discrimination between individuals with CP and neurotypical controls, and examined how these sensory variables relate to motor function, ADLs, and IADLs.

DETAILED DESCRIPTION:
Background: Sensory impairments are increasingly recognized as influential factors in the occupational performance of individuals with Cerebral Palsy (CP). Although prior studies have explored this relationship in children, evidence in young adults remains limited.

Objective: This study aimed to compare tactile sensitivity and discrimination in young adults with CP and neurotypical individuals, and to examine their association with motor-related variables relevant to occupational performance: muscle tone, grip strength, manual dexterity, Activities of Daily Living (ADLs), and Instrumental Activities of Daily Living (IADLs).

Methods: A multicenter cross-sectional study was conducted involving two groups of 36 participants aged 16-45 years. Sensory and motor variables were assessed using the Semmes-Weinstein Monofilaments, Two-Point Discrimination Test, Modified Ashworth Scale, Digital Dynamometer, Box and Block Test, Functional Independence Measure, and the Lawton and Brody Scale.

Conclusion: Findings highlight the relevance of sensory function in the occupational performance of young adults with CP. These results underscore the need for occupational therapy interventions that integrate sensory assessments and target sensory-motor integration to improve functional independence and participation.

ELIGIBILITY:
Inclusion Criteria:

* young people and adults with a medical diagnosis of CP, who had a motor condition of hemiparesis, diparesis, or tetraparesis;
* aged between 16 and 45 years
* had a minimum score of 19 on the Mini Mental State Examination cognitive assessment scale
* authorized their participation in the study by signing an informed consent form. In cases between the ages of 16 and 18 years, informed consent was signed by the participants and their parents or legal guardians

Exclusion Criteria:

* any peripheral nerve injury
* shoulder, elbow, wrist or hand injuries
* individuals whose mother tongue was neither Portuguese nor Spanish

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A multicenter cross-sectional study was conducted involving two groups of 36 participants aged 16-45 years.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Semmes-Weinstein monofilaments | 1 month
  This non-invasive technique assesses cutaneous sensory perception using nylon monofilaments of varying diameters that apply specific pressure forces. These forces range from 0.07 g (smallest) to 300 g (largest). In this study, monofilaments were applied to distinct areas innervated by different nerves: the distal phalanx of the first, second, and third fingers and the thenar eminence (median nerve), the fifth finger and hypothenar eminence (ulnar nerve), and the proximal phalanx of the first and second fingers on the dorsal side (radial nerve).
Two-point discrimination test | 1 month
  This test evaluates the ability to distinguish between two closely spaced pressure points on the skin, reflecting sensory acuity and receptor density. Distances typically range from 0 to 8 mm. Despite being widely used, standardization of pressure remains a challenge; a light, uniform pressure (10-15 g) is recommended. In this study, the same hand regions assessed with monofilaments were used. Proper simultaneous application was ensured to avoid perception bias.
Modified Ashworth Scale (MAS) | 1 month
  The MAS is widely used to evaluate muscle spasticity by measuring resistance to passive movement. The scale ranges from 0 (no tone increase) to 4 (severe rigidity), with the inclusion of score 1+ for greater sensitivity. In this study, assessments were performed on elbow and wrist flexor/extensor muscles, muscles involved in pronation/supination, and finger flexors/extensors. The scale helps quantify the degree of hypertonia, a common symptom in individuals with neurological conditions.
Digital dynamometer | 1 month
  Grip strength was measured using a handheld digital dynamometer, which quantifies isometric force output in kilograms. Testing was conducted with participants seated, shoulder adducted, elbow at 90º, forearm in neutral, and wrist extended 0º-30º. Both upper limbs were assessed. This measurement reflects overall upper limb strength and functional capacity, and is considered a reliable indicator of motor performance in clinical populations.
Box and Block Test | 1 month
  This test evaluates unilateral manual dexterity by counting the number of wooden blocks a participant can transfer from one side of a partitioned box to the other within 60 seconds. A 15-second practice trial was included to ensure familiarity with the procedure. It is a validated tool for individuals with neurological impairments and provides a quick, functional measure of hand coordination. Performance was assessed for both dominant and non-dominant hands.
Functional Independence Measure | 1 month
  The FIM assesses performance in Activities of Daily Living (ADLs) across two domains: motor (13 items) and cognitive/social (5 items). Each item is rated on a 7-point scale from total dependence (1) to complete independence (7), with a maximum total score of 126. It evaluates self-care, sphincter control, mobility, communication, and social cognition. This tool is widely used to determine the level of assistance required in daily life
Lawton and Brody Scale | 1 month
  This scale measures independence in Instrumental Activities of Daily Living (IADLs), such as using the telephone, managing medications and finances, shopping, cooking, and transportation. Scores range from 0 (dependent in all tasks) to 8 (independent in all tasks). It is particularly useful for evaluating more complex, community-based activities that are essential for independent living and is a standard tool in occupational therapy and geriatric assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Olalla Saiz Vazquez, Burgos, Burgos, Spain

IPD SHARING:
Plan to Share IPD: No
There is no data sharing plan for individual participant data (IPD) associated with this study. No IPD will be shared with other researchers.

REFERENCES:
- [Background] Kangas T. [Foot problems in diabetes]. Duodecim. 1981;97(12):872-8. No abstract available. Finnish. PMID 7297454
- [Background] Mesquita MA, Balbino EP, Albuquerque RS, Carmona CA, Okubo BT, Lorena SL, Montes CG, Soares EC. Ceftriaxone in the treatment of spontaneous bacterial peritonitis: ascitic fluid polymorphonuclear count response and short-term prognosis. Hepatogastroenterology. 1997 Sep-Oct;44(17):1276-80. PMID 9356840
- [Background] Bleyenheuft Y, Gordon AM. Precision grip control, sensory impairments and their interactions in children with hemiplegic cerebral palsy: a systematic review. Res Dev Disabil. 2013 Sep;34(9):3014-28. doi: 10.1016/j.ridd.2013.05.047. Epub 2013 Jun 29. PMID 23816634